CLINICAL TRIAL: NCT03837678
Title: Epithelioid Sarcoma Natural History Study
Status: Completed | Type: Observational
Sponsor: Epizyme, Inc. (Industry)
Collaborators: Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Other Study IDs: EZH-1001
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Epithelioid Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a multi-center, non-interventional retrospective medical records review. The study will involve identification of medical records of patients with confirmed locally advanced unresectable or metastatic ES, who initiated systemic therapy between January 1, 2000 and December 31, 2017.

Data for the chart review will be extracted retrospectively from eligible subjects' charts (electronic or paper). Information on prior surgical treatment and neoadjuvant/adjuvant therapies for ES will also be collected for ineligible subjects with a locally advanced or metastatic ES diagnosis who did not initiated systemic therapy. Data collected will be anonymized by the investigators and will not be traceable back to individual subjects by the sponsor (i.e., no protected health information [PHI] will be collected).

DETAILED DESCRIPTION:
The sampling period will span from January 1, 2000 to December 31, 2017. As the chart abstraction dates may be different across institutions due to contracting and other logistical issues, to avoid seeing biased outcomes that may be related to this type of heterogeneity, a consistent study end date will be imposed for all patients when conducting the analysis. Information before this study end date will be analyzed and used to conduct the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically confirmed, locally advanced unresectable or metastatic Epithelioid Sarcoma (ES) requiring systemic therapy during between January 1, 2000 and December 31, 2017. The date of the confirmed locally advanced unresectable or metastatic ES diagnosis is designated as the index date.
* Patients may have a date of ES diagnosis at an earlier stage prior to 2000 and still be eligible for the study
* Initiation of treatment with any systemic anti-cancer therapy for the treatment of their locally advanced unresectable or metastatic ES between January 1, 2000 and December 31, 2017
* At least 10 years of age at the index date

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of Epithelioid Sarcoma (ES) patients (approximately 70 to 100) from approximately five (5) academic centers (i.e., study sites) in the US. The sampling period will span from January 1, 2000 to December 31, 2017.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Real-word overall response rate (rwORR) | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to treatment failure
  Proportion of patients who have a documented radiological scan showing clinician-assessed complete response or less-than-complete response, of any duration, defined for each regimen and by line
Real-world duration of response (rwDOR) | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to treatment failure
  Duration of time between the first radiological scan showing documented tumor response (any time of response excluding SD) to first noted disease progression, or treatment discontinuation if no progression occurred. This is defined for each line of therapy and by regimen.

SECONDARY OUTCOMES:
Time from treatment initiation to treatment discontinuation | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to treatment failure
Time from treatment initiation to treatment failure | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to treatment failure
  Treatment failure is defined as discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death
Real-world disease control rate (rwDCR) | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to treatment failure
  Proportion of patients who have documented radiological scans showing clinician-assessed complete response or less-than-complete response, or stable disease lasting at least 32 weeks
Overall survival (OS) | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to death
Real-world time to tumor progression (rwTTP) | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 to tumor progression

OTHER OUTCOMES:
Safety Outcome: Occurrence of adverse events | Initiation of treatment with any systemic anti-cancer therapy for the treatment between January 1, 2000 and December 31, 2017 treatment modification or discontinuation
  Occurrence of adverse events resulting in treatment modification or discontinuation, or patient hospitalization, while on systemic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants. Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/